CLINICAL TRIAL: NCT01535248
Title: Echocardiographic Surveillance of Patients Undergoing Scheduled Endoscopic Retrograde Cholangiopancreatography for the Presence of Intracardiac Air Embolus
Brief Title: Echo Detection of Endoscopic Retrograde Cholangiopancreatography (ERCP) Air Embolus
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0238-11-FB
Record Dates: First submitted 2011-08-08; First posted 2012-02-17 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Air Embolism as A Complication of Medical Care
Keywords: ERCP; Transthoracic Echocardiography; Air Embolus; ERCP associated air embolus
MeSH Terms: conditions — Embolism, Air

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All ERCP Patients: All patients that will be approached for this study will be undergoing ERCP as part of their medical care.
  Interventions: Other: Transthoracic Echocardiography

INTERVENTIONS:
Other: Transthoracic Echocardiography — Patients undergoing ERCP will have surveillance with transthoracic echocardiography with exams occurring every 10 mins or more often if needed to evaluate for the presence of intra-cardiac air associated with ERCP insufflation.
  Other Names: Monitoring

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an endoscopy technique to visualize and evaluate the pancreatic and biliary systems. It has been reported that rare instances of air embolus have been found associated with the performance of an ERCP and many of these events are fatal. It is our proposal to use transthoracic echocardiography to continuously evaluate for the presence of intra-cardiac air secondary to ERCP venous air embolism and attempt to quantify the incidence of this complication and any potential patient factors that might increase the risk of this complication.

DETAILED DESCRIPTION:
Endoscopic Retrograde Cholangiopancreatography (ERCP) is commonly used in the diagnosis and treatment of biliary and pancreatic disease. There are case reports presented in the literature demonstrating adverse and often fatal events following air embolization associated with the performance of ERCP. The frequency of air embolus is extremely rare with the exact incidence unknown. In recent years the utilization of echocardiography to evaluate individuals with hemodynamic instability has led to the discovery of intracardiac air embolus seen in those individuals that demonstrated changes in either hemodynamic parameters or capnography values. There exists proposed mechanisms for the translocation of air from the foregut to the systemic venous circulation but not one of these mechanisms has yet been validated. Some proposed mechanisms include either through intrahepatic mechanisms where air crosses from the biliary tract to hepatic venules or potentially from the foregut into the portal vein and through shunt vessels into systemic venous circulation.

The exact frequency of air embolus is likely higher than the incidence of fatal or near-fatal complications reported in the literature. Individuals that had the best outcomes were usually intubated and had capnography to demonstrate a change suggestive of air embolus prior to significant hemodynamic changes.1 As this phenomenon has not previously been well described, it is possible that other patients suffer significant air embolus with myocardial or cerebral ischemic sequelae that were not recognized because echocardiography was not used as an early tool for evaluation of hemodynamically unstable patients. It is also possible that there are a number of patients that may suffer a venous air embolus from ERCP that is sub-clinical and therefore not causing enough change in cardiac function to alter either hemodynamic parameters or capnography values. The literature suggests that if a patient does not awake following ERCP, that imaging modalities, such as echocardiography be employed for evaluation.1 Understanding the frequency of this problem or which subgroups are at risk can further aid in the diagnosis and treatment of this complication.

Transthoracic echocardiography is a highly sensitive imaging modality and if adequate imaging windows can be obtained will demonstrate the presence of intracardiac air. The risk of performing the study on the patient is zero to very low. The potential risk of inaccurate interpretation should be avoided by the use of trained individuals in the acquisition and interpretation of transthoracic echocardiographic images.

The purpose of this study is to 1) identify individuals scheduled to undergo elective ERCP as part of their plan-of-care and perform transthoracic echocardiography for surveillance of intracardiac air embolus 2) record aspects of their past medical history that may potentially contribute to increased risk of systemic venous air embolus. This evaluation has not been presented in the literature and the primary end-point of this study would be to determine the frequency at which venous air embolus associated with ERCP occurs.

All individuals that meet inclusion criteria will be approached and consented in the pre-operative area prior to the planned procedure (ERCP). Their past medical history will be reviewed with the patient and special attention placed on particular co-morbid conditions that might be related to this phenomenon including but not limited to: portal hypertension, cirrhosis, portal vein thrombosis, and recent liver biopsy. The patient will then proceed to the procedure room as planned and while the patient is placed in the left lateral decubitus position and induced under anesthesia. An echocardiography-trained anesthesiologist will perform a transthoracic echocardiogram (TTE) concurrently while the gastroenterologist is performing the ERCP. We plan on conducting serial images at least every ten to fifteen minutes throughout the ERCP and more often as needed. At the conclusion of the procedure (ERCP) if there are no significant findings on TTE the patient will be returned to the supine position and taken to the recovery room. The written record of the TTE will then be entered into the study database within a separate research chart. In the event that the TTE shows the presence of intracardiac air embolus during the procedure the member of the study group performing the TTE will notify the endoscopist and anesthesia provider of the findings if the findings are significant enough to require a change in the patient's medical care. Reference to the algorithm will be made in each case and be available online if needed. Unless a moderate to severe embolic event occurs, the findings will not be communicated to the gastroenterologist so that he is blinded to the result maintained in the research chart. The purpose of this is to keep clinically insignificant emboli from being reported in the patient's medical record.

One of the key components of this evaluation is determining whether the presence of an air embolus has occurred and if so, has it had a negative effect on the function of the subject's cardiovascular system. Our proposed evaluation of the myocardium using transthoracic echocardiography includes evaluation of the left ventricle, right ventricle and pulmonary artery pressures. In the event there is hemodynamic instability as a result of impaired function of the right or left ventricle, an evaluation including measurements of the following parameters will assist in determination of the problem:

1. Right ventricular function, specifically tricuspid annular plane systolic excursion (TAPSE and the presence of hemodynamic changes.
2. Left ventricular function, specifically diastolic function, systolic function and myocardial performance index.
3. Pulmonary artery systolic pressure, via evaluation of the tricuspid regurgitant jet maximum velocity using the modified Bernoulli equation.
4. Presence of a new right-to-left intracardiac shunt or bowing of the intraatrial septum from right-to-left indicating a new increase in the right atrial pressure.
5. Significant changes in hemodynamic status that would indicate that the subject does not have effective filling and ejection of the left ventricle to support a perfusing blood pressure. This may manifest as hypotension and/or tachyarrhythmias on standard intraoperative monitoring.

As this protocol evaluates the frequency and degree of air embolization into the systemic venous system during the performance of endoscopic retrograde cholangiopancreatography (ERCP), the following four subgroups have been identified to help define the identification and treatment of subjects enrolled into IRB 238-11. Each category has a) criteria for the visual quantification of the air seen and b) the cardiac function and hemodynamic changes seen and finally c) the planned intervention if needed:

1. No air embolism:

   1. No visualized air emboli during the procedure.
   2. Subjects have no hemodynamic or myocardial changes attributable to the occurrence of venous air embolus.
   3. No changes would be made to the standard care of this research subject as a result of the absence of findings. Findings will be entered into the research chart.
2. Small air embolism:

   1. A small, but identifiable quantity of air visualized that does not form a large collection and does not obscure visualization of the far-field.
   2. Subjects have no changes in myocardial function and maintenance of hemodynamics.
   3. The subject would then undergo follow-up evaluation by a member of the study group at the conclusion of their normal post-op recovery period. No additional time would be required for evaluation and documentation of hemodynamic stability and follow-up echocardiography findings would be recorded in the research chart.
3. Moderate air embolism :

   1. Identifiable intracardiac air within the heart that obscures the far-field due to its size but does not cause a sharp demarcation at the blood/gas interface.
   2. Subjects have documented impairment of myocardial function and/or hemodynamics compared to baseline but do not require emergency resuscitation to correct.
   3. The subject would remain in the left lateral decubitus ("safe position" for individuals with suspected or confirmed venous air embolism) for four hours. Laboratory tests including cardiac enzymes may be obtained and a member of the study team will re-evaluate with transthoracic echocardiography. If baseline function and hemodynamics return, the subject concludes their recovery period as per normal circumstance for ERCP. In the event the subject has persistent intracardiac air, impaired myocardial function or hemodynamic instability, it would be recommended that the subject stay for observation with telemetry monitoring and further evaluation as needed.
4. Large air embolism:

   1. Identifiable intracardiac air which collects into a large enough bubble to cause sharp demarcation at the blood/gas interface and obscures the far-field.
   2. Left and/or right ventricular failure with hemodynamic collapse.
   3. The subject would require emergency resuscitation and ACLS protocol in addition to placement of invasive monitors for evaluation. Attempts to extract intracardiac air using central venous catheter will be made and as needed intubation with transfer to the ICU for further monitoring. Consultation for hyperbaric oxygen therapy would be pursued and all measures would be taken to recover hemodynamic function.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing ERCP as part of their medical care
* Subject will be of age 19 or older

Exclusion Criteria:

* Subject positioning for the ERCP is prone, thereby inhibiting the performance of the TTE
* Subject intolerance of the pressure of the TTE probe
* Subject body habitus interferes with obtaining adequate images to assess for intra-cardiac air

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Study Population will be all subjects who are scheduled to undergo ERCP and consent to participate in the protocol. No exclusions will be made based on gender or race to provide for a particular distribution, all subjects who would like to participate will be included.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-03-07; Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of ERCP associated air embolism | Participation will be for one day, during the time of the ERCP
  Patients who are scheduled for ERCP as part of their routine care will be assessed for the presence of air embolus, both clinically relevant (in the form of hemodynamic changes) and those situations where air is identified and does not appear to have a clinical effect. This is scheduled to occur over one day's time and only during the procedure are we planning on performing the echo for surveillance of air emboli.

SECONDARY OUTCOMES:
Risk Factors associated with ERCP air embolus | Participation will be for one day, during the time of the ERCP
  If it is found that there is a significant number of individuals that are found to have ERCP associated air embolus it would be a secondary goal to attempt to identify patient factors that might confer additional risk of air embolus to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas W Markin, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States